CLINICAL TRIAL: NCT00679874
Title: Characterization of the Cardiotoxic Effects of Chemotherapies With Anthracyclines and Trastuzumab for Breast Cancer by Contrast-enhanced Cardiovascular Magnetic Resonance Imaging (CMR).
Brief Title: Assessment of Cardiotoxicity After Chemotherapy for Breast Cancer by Cardio-vascular Magnetic Resonance (MR)
Acronym: Cardiotox
Status: Terminated | Type: Observational
Why Stopped: No subjects indentifiable
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Oliver Strohm, adunct Research Associate Professor, University of Calgary
Other Study IDs: Cardiotox_001
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Last update posted 2011-10-04 (Estimated); Status verified 2011-10

CONDITIONS: Breast Cancer
Keywords: Cardiovascular Magnetic Resonance Imaging; Cardiotoxicity; Anthracyclines; Trastuzumab; Breast cancer; Toxicity
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- I: Consecutive patients with first-time diagnosis of metastatic breast cancer undergoing chemotherapy with anthracyclines and/or trastuzumab.
  Interventions: Other: Cardio-vascular MRI

INTERVENTIONS:
Other: Cardio-vascular MRI — Contrast enhanced CMR studies at baseline, in the middle of chemotherapy and as follow-up

SUMMARY:
Consecutive patients with a first diagnosis of breast cancer will be identified at the Tom Baker Cancer Centre (TBCC) and included into the study, if they are going to receive chemotherapy with anthracyclines and / or Trastuzumab and do not have contra-indications for the CMR study. Besides the usual clinical care for these patients (e.g. blood samples before each cycle of chemotherapy; MUGA scans to follow cardiac size and function), the patients will undergo serial contrast-enhanced CMR studies (before, during and 9-12 months after completion of the chemotherapy); patients will be seen at an outpatient clinic in the Dept. of Cardiac Sciences / Heart Function Clinic for a clinical assessment (including ECG, additional blood test like Troponin-T, BNP, 6-minute-walk-test) and recommendations will be made to medical treatment in patients with evidence for heart failure.

Time points for the CMR and clinic assessments will be co-coordinated with regularly scheduled test by the TBCC to avoid unnecessary burden for the patients. The oncologists at the TBCC will be blinded to the results of the CMR studies and to laboratory results, unless the participating cardiologists identify a clinical need for communication.

Standardized CMR protocols will be employed and all interpretations will be blinded to the time course of the chemotherapy and cardiotoxic side effects.

We will test the hypothesis, whether CMR can be useful in patients with potentially cardiotoxic chemotherapy to:

* Identify patients at risk for the development of grade 2-4 cardiotoxic side effects as classified by the NCI guidelines (common toxicity criteria, 2001, 1-12)
* Identify imaging parameters to predict early or late Cardiotoxicity
* Provide additional clinical information to optimize medical treatment for heart failure

DETAILED DESCRIPTION:
Study Focus and Design:

Breast cancer is one of the leading cancers among white and African American women; its incidence has increased from one in 20 in 1960 to one in eight today ARMSTRONG 2000. In Canada alone, approximately 22,000 women are diagnosed each year with breast cancer and over 5,000 die from it VERMA 2007. Surgery, radiation therapy and/or chemotherapy are the most commonly used treatment options. Anthracyclines, especially doxorubicin, are a class of chemotherapeutic agents with efficacy against a variety of solid tumors, including breast cancer. Unfortunately, cardiotoxic effects occur with cumulative doses and limit the clinical use of doxorubicin. The incidence of heart failure is less than 5% at doses below 500 mg/m2, but increases to 18% with doses of 500 - 550 mg/m2 and exceeds 30% at doses of more than 600 mg/m2 1-5. Although several mechanism have been proposed for the cardiotoxic effects, little is known about prevention and effective treatment of this drug-induced cardiomyopathy.

The human epidermal growth factor receptor 2 (HER-2), also known as ErbB2, is a member of the group of transmembrane tyrosine kinases and is involved in the regulation of cell proliferation GSCHWIND2004. In mice with genetic defects in ErbB2, the ventricle fails to undergo trabeculation CRONE 2002; mice with reduced expression of HER-2 develop a dilated cardiomyopathy.

Approximately one quarter of patients with breast cancer have increased expression of HER-2, which is associated with a poorer prognosis including positive lymph nodes, decreased hormone receptor expression and high proliferative rates.

Trastuzumab (Herceptin) is a monoclonal antibody against the extracellular domain of HER-2 CARTER1992 and was approved for treatment of patients with HER-2 positive metastatic breast cancer in the 1990´s VOGEL 2002. Later, trastuzumab was approved for the use following anthracycline-based chemotherapies to decrease disease progression and to improve survival. The combination of anthracyclines and trastuzumab in the adjuvant setting reduced the risk of breast cancer relapse by 50% and the risk of death from breast cancer by 33% PICCARD 2005 und ROMOND 2005.

Despite the proven therapeutic benefits, trastuzumab shows cardiotoxic side effects in up to 25% of treated patients, especially if used in combination with doxorubicin. Approximately 5-10% of all patients treated with trastuzumab in the adjuvant setting develop (mostly asymptomatic) cardiac dysfunction and 1-3% develops severe and highly symptomatic heart failure with NYHA functional class III - IV CHIEN 2006. While both early (peaking 4 months post chemotherapy) and late (up to several years post exposure) cardiac toxicities leading to congestive heart failure have been described following administration of anthracycline-based chemotherapy, the pathophysiology of this toxicity, particularly in the late phase remains incompletely understood and several mechanism have been proposed; the interruption of the HER-2 signaling pathway in the heart seems to affect the ability of cardiomyocytes to grow, repair and survive. Studies in HER-2 knock-out mice have shown that a dilated cardiomyopathy develops following cardiac stress with anthracycline administration OZCELIK 2002. A direct toxic effect of the HER-2 blockade on the myocardial tissue level has been discussed, too OZCELIK 2002, trastuzumab seems to block anti-apoptotic signaling pathways, leading to cardiac dysfunction OZCELIK 2002.

An autopsy series of cancer patients having received anthracyclines demonstrated that 65% of patients with clinical CHF had microscopic evidence of drug toxicity, but that 35% did not 6. It may be difficult to distinguish anthracycline cardiac toxicity (ACT) from other causes using other currently available non-invasive modalities 3.

The trastuzumab-induced left ventricular dysfunction seems to reversible in the majority of cases, but little is known on the real-world effects of anthracyclines and trastuzumab on cardiac function during chemotherapy and shortly after.

CMR is the non-invasive gold standard in cardiac imaging for the assessment of cardiac function and also for the characterization of the myocardium and is used for the assessment of other acquired myocardial changes as myocarditis 7 and non-ischemic cardiomyopathies. Pilot studies have shown that CMR can detect even sub-clinical cardiotoxic effects in patients after anthracycline chemotherapy 8.

Our suggested study will prospectively include patients with a first diagnosis of breast cancer undergoing potentially cardiotoxic chemotherapy to identify the predictive value of several CMR-derived identifiers for cardiotoxicity and to evaluate an individually adjusted follow-up by cardiologists during and after the chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* First-time diagnosis of breast cancer
* Planned chemotherapy with anthracyclines and / or Trastuzumab
* Ability to give informed consent

Exclusion Criteria:

* Contra-indications for CMR study (e.g. implanted pacemaker / ICD; severe renal impairment (GFR< 35 ml/min); severe claustrophobia)
* Previous history of non-ischemic cardiomyopathies or myocardial inflammation
* Inability to give informed consent
* Concomitant drug abuse (e.g. cocaine)
* Expected life expectancy < 6 months

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients with a first diagnosis of breast cancer will be identified at the Tom Baker Cancer Centre (TBCC) and included into the study, if they are going to receive chemotherapy with anthracyclines and / or Trastuzumab and do not have contra-indications for the CMR study.
Sampling Method: Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2008-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Drop in ejection fraction of 10% as compared to baseline | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Strohm, MD, FESC, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Dept. of Cardiac Sciences and Tom Baker Cancer Centre, Calgary, Alberta, Canada

REFERENCES:
- [Background] Nathan DM. Rosiglitazone and cardiotoxicity--weighing the evidence. N Engl J Med. 2007 Jul 5;357(1):64-6. doi: 10.1056/NEJMe078117. Epub 2007 Jun 5. No abstract available. PMID 17551161
- [Background] McArthur HL, Chia S. Cardiotoxicity of trastuzumab in clinical practice. N Engl J Med. 2007 Jul 5;357(1):94-5. doi: 10.1056/NEJMc070065. No abstract available. PMID 17611218
- [Background] Wassmuth R, Lentzsch S, Erdbruegger U, Schulz-Menger J, Doerken B, Dietz R, Friedrich MG. Subclinical cardiotoxic effects of anthracyclines as assessed by magnetic resonance imaging-a pilot study. Am Heart J. 2001 Jun;141(6):1007-13. doi: 10.1067/mhj.2001.115436. PMID 11376317
- [Background] Friedrich MG, Strohm O, Schulz-Menger J, Marciniak H, Luft FC, Dietz R. Contrast media-enhanced magnetic resonance imaging visualizes myocardial changes in the course of viral myocarditis. Circulation. 1998 May 12;97(18):1802-9. doi: 10.1161/01.cir.97.18.1802. PMID 9603535